CLINICAL TRIAL: NCT00736697
Title: An Open-Label, Randomized, Single-Dose, Parallel-Group Study to Determine the Effect of a High-Fat Meal on the Relative Bioavailability and Pharmacokinetics of a Single Dose of Moxidectin Administered Orally to Healthy Subjects
Brief Title: Study Evaluating The Effect Of High-Fat Meal On Bioavailability And Pharmacokinetics Of Single Dose Of Moxidectin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 3110A1-1005
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Last update posted 2011-02-15 (Estimated); Status verified 2011-02

CONDITIONS: Infection
MeSH Terms: conditions — Infections | interventions — moxidectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: moxidectin

INTERVENTIONS:
Drug: moxidectin

SUMMARY:
The primary objective of this study is to assess the effect of a high-fat meal (breakfast) on the concentrations of moxidectin measured in the blood after a single oral administration in healthy subjects.

ELIGIBILITY:
Inclusion Criteria

* Men or women of non childbearing potential aged 18 to 50 years inclusive at screening.
* Body mass index (BMI) in the range of 18.0 to 30.0 kg/m2 and body weight greater than or equal to 50 kg.

Exclusion criteria

* Any clinical important deviation from normal limits in physical examination findings, vital sign measurements, electrocardiograms or clinical laboratory test results.
* Presence or history of any disorder that may prevent the successful completion of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2008-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Blood samples | 4 months

SECONDARY OUTCOMES:
Electrocardiograms | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Poitiers, France